CLINICAL TRIAL: NCT03752853
Title: Biological Correlates of an Internet-based Psychological Intervention for Depression
Brief Title: Stress Systems and Psychotherapy in Depression
Acronym: Bio-COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Responsible Party: Principal Investigator, Dr. Sarah Schumacher, Principal Investigator, Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stress_DEP
Record Dates: First submitted 2018-11-13; First posted 2018-11-26 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Episode
Keywords: major depressive episode; cortisol; alpha-amylase; psychotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCBT for depression - behavioral activation first (BAF) (Experimental): internet-based intervention for mild to moderate depression: patients receive behavioral activation first, followed by cognitive restructuring
  Interventions: Behavioral: internet-based intervention for mild to moderate depression
- iCBT for depression - cognitive restructuring first (CRF) (Experimental): internet-based intervention for mild to moderate depression: patients receive cognitive restructuring first, followed by behavioral activation
  Interventions: Behavioral: internet-based intervention for mild to moderate depression

INTERVENTIONS:
Behavioral: internet-based intervention for mild to moderate depression — The six-weeks, therapist-guided, internet-based intervention for depression includes expressive writing tasks and further consists of key elements of cognitive behavioral therapy (CBT) for depression. In seven consecutive modules, patients receive psychoeducation and instructions for weekly tasks, and an individualized feedback letter of their therapist after each module. The intervention is effective in reducing depressive symptoms (Zagorscak et al., 2018). In the current study, patients will be randomly assigned to two different conditions with varying orders of modules: 1. patients will receive two modules (module 3 and 4) of behavioral activation, followed by two modules (modules 5 and 6) of cognitive restructuring; 2. patients will receive two modules (module 3 and 4) of cognitive restructuring, followed by two modules (modules 5 and 6) of behavioral activation. All other modules (1, 2 and 7) will be identical across conditions.

SUMMARY:
Dysregulation of the hypothalamus-pituitary-adrenal (HPA) axis as well as maladaptive activation of the autonomic nervous system (ANS) are discussed as relevant factors in the development of a major depressive episode and as a correlate of its clinical manifestation. Preliminary evidence suggests that the hypercortisolaemic pattern in a subgroup of depressed patients may predict non-responses to psychotherapeutic treatment. At the same time, it is conceivable that disorder-related alterations in HPA axis and ANS regulation change in response to effective treatment, such as cognitive behavioural therapy (CBT), and that those changes could parallel changes in depressive symptoms. Identifying such associations may shed light on biological and psychological mechanisms of action underlying successful treatment.

However, so far, no studies have investigated depressed patients with regard to dysregulation in both stress systems, HPA axis and ANS, before psychotherapeutic treatment, nor have changes in functioning of both systems been inspected in response to treatment. Moreover, a detailed investigation of depressive symptom trajectories over the course of treatment and its associations with changes in HPA axis and ANS regulation is lacking. It can be speculated that specific techniques of the treatment, e.g., typical CBT elements, such as behavioural activation or cognitive restructuring, might particularly be associated with changes in HPA axis and ANS regulation.

The main aims of this project are to investigate:

1. whether diurnal salivary cortisol and alpha-amylase as well as hair cortisol concentrations change from pre- to post-intervention in treatment responders compared to non-responders;
2. whether diurnal salivary cortisol and alpha-amylase concentrations change from pre- to mid-intervention and from mid- to post-intervention in treatment responders compared to non-responders;
3. whether changes in diurnal salivary cortisol, alpha-amylase and hair cortisol concentrations are significantly correlated with changes in depressive symptoms;
4. whether concentrations of diurnal salivary cortisol and alpha-amylase as well as hair cortisol at pre-treatment predict future treatment response (i.e., on a psychological level).

   On an exploratory level, it will be investigated:
5. which elements of a CBT intervention for depression (behavioural activation vs. cognitive restructuring) are associated with changes in diurnal salivary cortisol and alpha-amylase concentrations.

It is hypothesised:

1. that pre- to post-intervention decreases in diurnal salivary cortisol and alpha-amylase as well as hair cortisol concentrations will be more pronounced in responders compared to non-responders.
2. that pre- to mid-intervention and mid- to post-intervention decreases in diurnal salivary cortisol and alpha-amylase will be more pronounced in responders compared to non-responders.
3. that changes in depressive symptoms will significantly correlate with changes in diurnal cortisol and diurnal alpha-amylase as well as hair cortisol concentrations.
4. that pre-intervention diurnal salivary cortisol and alpha-amylase as well as hair cortisol concentrations will be higher in future non-responders, compared to responders.

DETAILED DESCRIPTION:
Recruitment:

Patients will be recruited from an ongoing project providing an internet-based cognitive behavioral intervention for patients suffering from mild to moderate depression.

Protocol:

In this study, a total of N=42 patients fulfilling criteria for a current major depressive episode will undergo a 6-week internet-based cognitive behavioural intervention which consists of seven consecutive modules. Diurnal (salivary) and hair cortisol as well as diurnal (salivary) alpha-amylase will be assessed immediately before and after treatment, and at mid-treatment (i.e., after four of seven modules). Saliva samples (six samples per day) will be collected over two consecutive days. One hair sample will be obtained at pre- and post-intervention assessments respectively.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive episode (F32.0, F32.1, F33.0, F33.1)
* Agreement to participate in the study
* At least 18 years of age

Exclusion Criteria:

* Diagnosis of schizophrenia, schizotypal and delusional disorders (F20-F29)
* Acute suicidal patients
* Acute manic episode
* Substance related abuse or addiction
* Pregnancy or lactation
* Chronic somatic diseases
* Severe somatic diseases (e.g., endocrinological, neurological, autoimmune diseases)
* Glucocorticoid medication intake during the last six months
* Concurrent psychotherapeutic treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
Changes in salivary cortisol concentration | pre-intervention, mid-intervention (after an average of three weeks), post-intervention (after an average of six weeks)
  Changes in diurnal profiles (six time points: awakening, +30 min., 11am, 2 pm, 6pm, 9pm) of salivary cortisol concentration (nmol/l), measured on two consecutive days, at mid-intervention and post-intervention in responders compared to non-responders to the psychological intervention (assessed by Patient Health Questionnaire (PHQ-9))
Differences in salivary cortisol concentration | pre-intervention
  Differences in diurnal profiles (six time points: awakening, +30 min., 11am, 2 pm, 6pm, 9pm) of cortisol concentration (nmol/l), measured on two consecutive days, at pre-intervention in responders compared to non-responders to the psychological intervention (assessed by PHQ-9)
Changes in salivary alpha-amylase concentration | pre-intervention, mid-intervention (after an average of three weeks), post-intervention (after an average of six weeks)
  Changes in diurnal profiles (six time points: awakening, +30 min., 11am, 2 pm, 6pm, 9pm) of salivary alpha-amylase concentration (U/ml), measured on two consecutive days, at mid-intervention and post-intervention in responders compared to non-responders to the psychological intervention (assessed by Patient Health Questionnaire (PHQ-9))
Differences in salivary alpha-amylase concentration | pre-intervention
  Differences in diurnal profiles (six time points: awakening, +30 min., 11am, 2 pm, 6pm, 9pm) of salivary alpha-amylase concentration (U/ml), measured on two consecutive days, at pre-intervention in responders compared to non-responders to the psychological intervention (assessed by PHQ-9)
Changes in hair cortisol concentration | pre-intervention, post-intervention (after an average of six weeks)
  Changes in hair cortisol concentrations (nmol/l) at post-intervention in responders compared to non-responders to the psychological intervention (assessed by Patient Health Questionnaire (PHQ-9))
Differences in hair cortisol concentration | pre-intervention
  Differences in hair cortisol concentrations (nmol/l) at pre-intervention in responders compared to non-responders to the psychological intervention (assessed by PHQ-9)

SECONDARY OUTCOMES:
Sleep quality (self-report) | pre-intervention, mid-intervention (after an average of three weeks), post-intervention (after an average of six weeks)
  Changes in Pittsburgh Sleep Quality Index (PSQI); scale ranges from 0 to 21
Chronic stress (self-report) | pre-intervention, mid-intervention (after an average of three weeks), post-intervention (after an average of six weeks)
  Changes in Trier Inventory for the assessment of chronic stress - TICS (Trier Inventar zum chronischen Stress), scale ranges from 0 to 48
Cognitive biases (self-report) | pre-intervention, mid-intervention (after an average of three weeks), post-intervention (after an average of six weeks)
  Changes in Cognitive Styles Assessment (COSTA-21); scale ranges from 0 to 5 per item

CONTACTS AND LOCATIONS:
Locations (1):
- Freie Universitaet Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zagorscak P, Heinrich M, Sommer D, Wagner B, Knaevelsrud C. Benefits of Individualized Feedback in Internet-Based Interventions for Depression: A Randomized Controlled Trial. Psychother Psychosom. 2018;87(1):32-45. doi: 10.1159/000481515. Epub 2018 Jan 6. PMID 29306945